CLINICAL TRIAL: NCT06316999
Title: Utility of Intestinal Ultrasound as a Diagnostic Tool for the Evaluation of Pouchitis and Other Outcomes After Ileal Pouch-Anal Anastomosis: A Prospective Pilot Study
Brief Title: Intestinal Ultrasound for the Evaluation of Pouchitis and Other Outcomes After Ileal Pouch-Anal Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Darrell S. Pardi, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-012169
Record Dates: First submitted 2024-02-28; First posted 2024-03-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis; Pouchitis
Keywords: Ileal Pouch Anal Anastomosis
MeSH Terms: conditions — Colitis, Ulcerative; Pouchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with Pouchitis (Other): Transabdominal and transperineal ultrasounds of the pouch will be performed by an experienced sonographer for each patient and interpreted by a board-certified radiologist specializing in IUS.
  Interventions: Diagnostic Test: Intestinal Ultrasound

INTERVENTIONS:
Diagnostic Test: Intestinal Ultrasound — Transabdominal and trans perineal ultrasound of the pouch

SUMMARY:
Intestinal ultrasound (IUS) has been studied in the evaluation of inflammatory bowel disease (IBD) and is increasingly used as a non-invasive, easy to use, cost-effective tool for point-of-care to assess disease activity and more recently to predict response to treatment. However, there is a paucity of data on the use of IUS specifically for ulcerative colitis (UC) patients with an ileal pouch-anal anastomosis (IPAA).

DETAILED DESCRIPTION:
AIMS:

1. Establish normal sonographic parameters in patients with an IPAA and normal pouch function.
2. Evaluate the feasibility of IUS for diagnosing pouchitis and other outcomes and compare its performance with the current gold standard of pouchoscopy with biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Diagnosis of ulcerative colitis (UC)
* Status post ileal pouch anal anastomosis IPAA (completed all stages)

Exclusion Criteria:

* Pediatric patients
* Indeterminate colitis
* Status post IPAA for familial adenomatous polyposis (FAP)
* BMI > 30 kg/m2
* Pregnant
* Decompensated Cirrhosis
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of intestinal ultrasound (IUS) for pouchitis | through study completion, an average of 1 year
  compared to gold standard of pouchoscopy with biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Pardi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayoclinic.org/